CLINICAL TRIAL: NCT01461044
Title: An Ambispective, Non Interventional Study of 2 Cohorts (Triple Negative or HR+) of Patients With HER2- Metastatic or Locally Advanced Breast Cancer Treated With Avastin® (Bevacizumab) 1st Line for at Least 12 Months and Without Progression for at Least 12 Months.
Brief Title: An Observational Study of Avastin (Bevacizumab) in Patients With HER2-metastatic or Locally Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27760
Record Dates: First submitted 2011-10-24; First posted 2011-10-27 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the safety and efficacy of triple negative or HR+ patients with HER2-metastatic or locally advanced breast cancer treated with Avastin (bevacizumab) as first line therapy for at least 12 months and without disease progression for at least 12 months. Data will be collected retrospectively (from the diagnosis to the inclusion in the study) and for 18 months from study start.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* HER2-metastatic breast cancer or locally advanced breast cancer
* Patients with Avastin as first line therapy administered for at least 12 months
* Patients without disease progression after the beginning of Avastin treatment for at least 12 months

Exclusion Criteria:

* Patients not willing to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (triple negative or HR+) with HER2- metastatic or locally advanced breast cancer, treated with Avastin 1st line for at least 12 months and without progression for at least 12 months.
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (66):
- France (66):
  - Aix-en-Provence
  - Ajaccio
  - Amiens
  - Antony
  - Arras
  - Bastia
  - Bayonne
  - Beauvais
  - Besançon
  - Béziers
  - Bobigny
  - Bordeaux
  - Boulogne-Billancourt
  - Bourg-en-Bresse
  - Brest
  - Caen
  - Chambéry
  - Châteauroux
  - Cherbourg Octeville
  - Clermont-Ferrand
  - Créteil
  - Dax
  - Dijon
  - Eaubonne
  - Évreux
  - Grenoble
  - La Chaussée-Saint-Victor
  - La Roche-sur-Yon
  - La Tronche
  - Le Coudray
  - Lille
  - Limoges
  - Longjumeau
  - Lorient
  - Lormont
  - Lyon
  - Marseille
  - Metz
  - Montivilliers
  - Mougins
  - Nancy
  - Narbonne
  - Nice
  - Osny
  - Paris
  - Périgueux
  - Reims
  - Romans-sur-Isère
  - Rouen
  - Saint-Brieuc
  - Saint-Cloud
  - Saint-Germain-en-Laye
  - Saint-Grégoire
  - Saint-Jean
  - Saint-Michel-sur-Orge
  - Saint-Priest-en-Jarez
  - Senlis
  - Soyaux
  - Strasbourg
  - Toulon
  - Toulouse
  - Troyes
  - Valence
  - Vannes
  - Verdun
  - Villejuif

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 228 participants were included but 1 participant did not fulfill the inclusion criteria, therefore not included in the analysis. Inclusion (baseline) here was the time after the retrospective phase and at the start of prospective phase.
Groups:
- Bevacizumab: Hormone Receptor-Positive (HR+) Breast Cancer: Participants with human epidermal growth factor receptor 2 negative (HER2-) metastatic or locally advanced HR+ breast cancer, who received first-line bevacizumab in combination with chemotherapy for greater than or equal to (>=) 12 months and without disease progression for at least 12 months were included. Retrospective data were collected till inclusion in the study. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months. Bevacizumab treatment considering retrospectively and prospectively was approximately 61 months.
- Bevacizumab: Triple Negative (TN) Breast Cancer: Participants with HER2- metastatic or locally advanced TN breast cancer, who received first-line bevacizumab in combination with chemotherapy for >=12 months and without disease progression for at least 12 months were included. Retrospective data were collected till inclusion in the study. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months. Bevacizumab treatment considering retrospectively and prospectively was approximately 61 months.
Period: Overall Study
Arm/Group | Bevacizumab: Hormone Receptor-Positive (HR+) Breast Cancer | Bevacizumab: Triple Negative (TN) Breast Cancer
Started | 150 | 77
Participants Alive at Inclusion | 127 | 58
Completed | 80 | 37
Not Completed | 70 | 40
Not completed — Death | 58 | 35
Not completed — Lost to Follow-up | 12 | 5

BASELINE CHARACTERISTICS:
Population: Efficacy population included all participants who did not violate any inclusion or exclusion.
Groups:
- Bevacizumab: HR+ Breast Cancer: Participants with HER2- metastatic or locally advanced HR+ breast cancer, who received first-line bevacizumab in combination with chemotherapy for >=12 months and without disease progression for at least 12 months were included. Retrospective data were collected till inclusion in the study. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months. Bevacizumab treatment considering retrospectively and prospectively was approximately 61 months.
- Bevacizumab: TN Breast Cancer: Participants with HER2- metastatic or locally advanced TN breast cancer, who received first-line bevacizumab in combination with chemotherapy for >=12 months and without disease progression for at least 12 months were included. Retrospective data were collected till inclusion in the study. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months. Bevacizumab treatment considering retrospectively and prospectively was approximately 61 months.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer | Total
Number analyzed (Participants) | 135 | 67 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (12.0) | 55.6 (10.3) | 55.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 67 | 202
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Disease-Free for at Least 12 Months After Initial Diagnosis
Description: Disease free interval was expressed in months: (Date of diagnosis of metastatic disease - Date of initial diagnosis + 1) / 30.4375. Percentage of participants who were disease-free for at least 12 months were reported.
Time Frame: From initial diagnosis to the diagnosis of metastatic disease (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 134 | 67
percentage of participants | 73.1 [65.1 to 79.9] | 80.6 [69.6 to 88.3]

2. Secondary Outcome: Percentage of Participants With a Best Overall Response (BOR) of Confirmed Complete Response (CR) or Partial Response (PR)
Description: Objective tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR was defined as the disappearance of all target and non-target lesions, and confirmed PR was defined as at least at 30% decrease in the sum of the longest diameters of target lesions. Response was to be confirmed at follow-up assessment completed within 4 weeks of the first documented response. Inclusion (baseline) here was the time after the retrospective phase and at the start of prospective phase.
Time Frame: From first administration of bevacizumab to inclusion in the study (up to a maximum of 42.8 months , assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 131 | 59
percentage of participants
  CR | 28.2 [21.2 to 36.5] | 33.9 [23.1 to 46.6]
  PR | 58.0 [49.5 to 66.1] | 45.8 [33.7 to 58.3]

3. Secondary Outcome: Percentage of Participants With Disease Progression or Death
Description: Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death"). PD was defined as the appearance of new lesion(s) or at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum obtained at Screening or during treatment.
Time Frame: as for outcome 2
Population: Efficacy population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
percentage of participants | 79.3 | 80.6

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival was defined as the time from first dose of bevacizumab to documented PD or death from any cause, whichever occurred first. PD was defined as the appearance of new lesion(s) or at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum obtained at Screening or during treatment. Inclusion (baseline) here was the time after the retrospective phase and at the start of prospective phase.
Time Frame: From first administration of bevacizumab to inclusion in the study (up to a maximum of 42.8 months, assessed retrospectively at Baseline)
Population: Efficacy population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
months | 25.3 [22.4 to 31.1] | 21.2 [19.1 to 25.4]

5. Secondary Outcome: Time to Progression
Description: Objective tumor response was assessed using RECIST. PD was defined as the appearance of new lesion(s) or at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum obtained at Screening or during treatment. Participants who withdrew from the study early for insufficient therapeutic response without tumor assessment for PD were also included within the definition of PD. Time to progression was defined as the time from treatment start to PD. Participants who did not experience PD were censored from the last tumor assessment. Time to progression was estimated using Kaplan-Meier and expressed in months. Inclusion (baseline) here was the time after the retrospective phase and at the start of prospective phase.
Time Frame: as for outcome 4
Population: Efficacy population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
months | 25.3 [22.4 to 31.8] | 21.2 [19.1 to 25.4]

6. Secondary Outcome: Percentage of Participants With Death
Description: Overall survival (OS) was defined as the time between the first administration of bevacizumab and death from any cause and participants still alive at the end of the study were censored at the last consultation or last contact date.
Time Frame: From the first administration of bevacizumab to death from any cause (up to a maximum of 60.8 months including retrospective and prospective treatment)
Population: Efficacy population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
percentage of participants | 37.8 | 41.8

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the first administration of bevacizumab and death from any cause and participants still alive at the end of the study were censored at the last consultation or last contact date.
Time Frame: as for outcome 6
Population: Efficacy population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
months | 57.2 [50.7 to NA] — The upper limit of confidence interval (CI) was not estimable because more than 50% of participants were censored. | 49.4 [39.8 to NA] — The upper limit of CI was not estimable because more than 50% of participants were censored.

8. Primary Outcome: Percentage of Participants Who Were Disease-Free for at Least 24 Months After Initial Diagnosis
Description: Disease free interval was expressed in months: (Date of diagnosis of metastatic disease - Date of initial diagnosis + 1) / 30.4375. Percentage of participants who were disease-free for at least 24 months were reported.
Time Frame: as for outcome 1
Population: Efficacy population. Here number of participants analyzed were those who were available for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 134 | 67
percentage of participants | 68.7 [60.4 to 75.9] | 56.7 [44.8 to 67.9]

9. Primary Outcome: Disease-Free Interval
Description: Disease free interval was expressed in months: (Date of diagnosis of metastatic disease - Date of initial diagnosis + 1) / 30.4375. Disease free interval was observed retrospectively and assessed at inclusion period or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: as for outcome 1
Population: Efficacy population. Here number of participants analyzed were those who were available for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 134 | 67
months | 51.0 [0 to 259] | 28.0 [0 to 257]

10. Primary Outcome: Mean Age at the Time of Local or Metastatic Progression
Description: Time of local or metastatic progression is the time of advanced or metastatic diagnosis which was assessed at inclusion or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population.
Measure: Mean (Standard Deviation); unit: years
Groups:
- Bevacizumab: TN Breast Cancer: Participants with HER2- metastatic or locally advanced TN breast cancer, who received first-line bevacizumab in combination with chemotherapy for >=12 months and without disease progression for at least 12 months were included. Retrospective data collected till inclusion in the study. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months. Bevacizumab treatment considering retrospectively and prospectively was approximately 61 months.
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
years | 54.5 (11.8) | 55.5 (10.4)

11. Primary Outcome: Percentage of Participants With Menopausal Status at the Time of Local or Metastatic Progression
Description: Menopausal status included premenopausal and menopausal. Time of local or metastatic progression is the time of advanced or metastatic diagnosis which was assessed at inclusion or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the evaluation of menopausal status.
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab: HR+ Breast Cancer: Participants with HER2- metastatic or locally advanced HR+ breast cancer, who received first-line bevacizumab in combination with chemotherapy for >=12 months and without disease progression for at least 12 months were included. Retrospective data of participants with HR+ cancer, receiving first-line bevacizumab in combination with chemotherapy for at least 12 months, were collected till inclusion in the study. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months. Bevacizumab treatment considering retrospectively and prospectively was approximately 61 months.
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 117 | 59
percentage of participants
  Premenopausal | 31.6 | 18.6
  Menopausal | 68.4 | 81.4

12. Primary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) at the Time of Local or Metastatic Progression
Description: ECOG-PS measured on-therapy (time between first dose and last dose date with a 30-day lag) assessed participant's performance status on a 5 point scale: 0 equals (=) fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, but ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50 percentage [%] of waking hours [h]), capable of all self care, but unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hours; 4= completely disabled, cannot carry on any selfcare, totally confined to bed or chair and 5=Dead. Only participants that reported in any of the specified scale was reported. Time of local or metastatic progression is the time of advanced or metastatic diagnosis which was assessed at inclusion or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the evaluation of ECOG PS.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 122 | 53
percentage of participants
  0 | 46.7 | 54.7
  1 | 43.4 | 37.7
  2 | 9.0 | 7.5
  3 | 0.8 | 0.0

13. Primary Outcome: Mean Body Weight at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the evaluation of body weight.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 131 | 66
kilograms | 66.8 (13.3) | 66.2 (11.1)

14. Primary Outcome: Mean Height at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the evaluation of height.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 128 | 63
centimeters | 161.7 (5.9) | 164.1 (5.6)

15. Primary Outcome: Mean Body Mass Index (BMI) at the Time of Local or Metastatic Progression
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2). Time of local or metastatic progression is the time of advanced or metastatic diagnosis which was assessed at inclusion or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the evaluation of BMI which was measured in kg/m^2.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 128 | 63
kg/m^2 | 25.6 (4.9) | 24.7 (4.2)

16. Primary Outcome: Percentage of Participants With Breast Cancer (BRCA) Mutation at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the evaluation of BRCA mutation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 130 | 65
percentage of participants | 1.5 | 4.6

17. Primary Outcome: Percentage of Participants With Metastatic Disease at Identified Metastatic Sites at the Time of Local or Metastatic Progression
Description: Metastatic diseases were identified at bone, lung, liver, central nervous system, soft tissue, lymph nodes, skin, pleura and other sites. Time of local or metastatic progression is the time of advanced or metastatic diagnosis which was assessed at inclusion or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
percentage of participants
  Bone | 63.7 [55.3 to 71.3] | 46.3 [34.9 to 58.1]
  Lung | 34.1 [26.6 to 42.4] | 29.9 [20.2 to 41.7]
  Liver | 35.6 [28.0 to 43.9] | 17.9 [10.6 to 28.7]
  Central nervous system | 2.2 [0.5 to 6.4] | 4.5 [0.9 to 12.5]
  Soft tissue | 10.4 [6.3 to 16.7] | 14.9 [8.3 to 25.3]
  Lymph nodes | 11.9 [7.4 to 18.4] | 28.4 [19.0 to 40.1]
  Skin | 5.2 [2.1 to 10.4] | 4.5 [0.9 to 12.5]
  Pleura | 6.7 [3.1 to 12.3] | 7.5 [2.5 to 16.6]
  Other | 8.1 [4.1 to 14.1] | 7.5 [2.5 to 16.6]

18. Secondary Outcome: Duration of Bevacizumab as First Line Treatment
Time Frame: From start of bevacizumab until 18 months after inclusion (up to a maximum of 60.8 months including retrospective and prospective treatment)
Population: Efficacy population.
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
months | 21.2 [12.0 to 60.8] | 18.6 [11.6 to 46.7]

19. Secondary Outcome: Percentage of Participants With Temporary Discontinuation
Time Frame: as for outcome 18
Population: Efficacy population. Here number of participants were those who were temporary discontinued.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
percentage of participants | 28.1 | 29.9

20. Secondary Outcome: Percentage of Participants With Reasons for Temporary Discontinuation
Time Frame: as for outcome 18
Population: Efficacy population. Here number of participants were those who were temporary discontinued.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 38 | 20
percentage of participants
  Adverse Event | 34.2 | 35.0
  Surgery | 34.2 | 45.0
  Participant's or Investigator's Decision | 15.8 | 20.0
  Unspecified | 21.1 | 10.0

21. Secondary Outcome: Percentage of Participants With Definitive Discontinuation
Time Frame: as for outcome 18
Population: Efficacy population. Here number of participants were those who were temporary discontinued.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
percentage of participants | 75.6 | 88.1

22. Secondary Outcome: Percentage of Participants With Reasons for Definitive Discontinuation
Time Frame: as for outcome 18
Population: Efficacy population. Here number of participants were those who were definitive discontinued.
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab: HR+ Breast Cancer: Participants with HR+ cancer, who received first-line bevacizumab in combination with chemotherapy for >=12 months and without disease progression for at least 12 months were included. Retrospective data of participants with HR+ cancer, receiving first-line bevacizumab in combination with chemotherapy for at least 12 months, were collected till inclusion in the study. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months.
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 102 | 59
percentage of participants
  Progressive disease | 54.9 | 58.6
  Adverse event | 24.5 | 24.1
  Participant's or Investigator's decision | 16.7 | 15.5
  Unspecified | 3.9 | 1.7

23. Primary Outcome: Percentage of Participants Classified Based on Number of Metastatic Sites at the Time of Local or Metastatic Progression
Description: Percentage of participants that reported metastatic disease in less than or equal to (<=) 3 sites or greater than (>) 3 sites were assessed. Time of local or metastatic progression is the time of advanced or metastatic diagnosis which was assessed at inclusion or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the evaluation of metastatic sites.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 134 | 66
percentage of participants
  <=3 | 56.7 [48.3 to 64.8] | 71.2 [59.4 to 80.7]
  >3 | 43.3 [35.2 to 51.7] | 28.8 [19.3 to 40.6]

24. Primary Outcome: Percentage of Participants With Visceral Involvement at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
percentage of participants | 64.4 [56.1 to 72.0] | 43.3 [32.1 to 55.2]

25. Primary Outcome: Percentage of Participants With Estrogen Receptors (ER) at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 90 | 43
percentage of participants
  ER+ | 92.2 | 0
  ER- | 4.4 | 93.0
  Unknown | 3.3 | 7.0

26. Primary Outcome: Percentage of Participants With Progesterone Receptors (PR) at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 90 | 43
percentage of participants
  PR+ | 64.4 | 0
  PR- | 31.1 | 93.0
  Unknown | 4.4 | 7.0

27. Primary Outcome: Percentage of Participants With Cross Results for Both ER and PR at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 86 | 40
percentage of participants
  ER+/PR+ | 64.0 | 0
  ER+/PR- | 31.4 | 0
  ER-/PR+ | 3.5 | 0
  ER-/PR- | 1.2 | 100

28. Primary Outcome: Percentage of Participants With HR Status at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 87 | 40
percentage of participants
  HR+ | 98.9 | 0
  HR- | 1.1 | 100

29. Primary Outcome: Percentage of Participants With Negative HER2 Status at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 91 | 40
percentage of participants | 100 | 100

30. Primary Outcome: Percentage of Participants With Mitotic Index (MI) at the Time of Local or Metastatic Progression
Description: MI is an indirect measure of cell proliferation that has been demonstrated to be a strong predictor of outcome for several human and canine cancers. Percentage of participants that reported a low, intermediate, high and unknown indices were included. Time of local or metastatic progression is the time of advanced or metastatic diagnosis which was assessed at inclusion or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 79 | 40
percentage of participants
  Low | 22.8 | 7.5
  Intermediate | 5.1 | 5.0
  High | 3.8 | 17.5
  Unknown | 68.4 | 70.0

31. Primary Outcome: Percentage of Participants With Ki67 (MiB1) at the Time of Local or Metastatic Progression
Description: The Ki67 (MiB1) a prognostic marker, is used to evaluate the proliferative activity of breast cancer. Percentage of participants with < or >=10% and unknown were reported. Time of local or metastatic progression is the time of advanced or metastatic diagnosis which was assessed at inclusion or baseline (the time after the retrospective phase and at the start of prospective phase).
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 80 | 38
percentage of participants
  <10% | 3.8 | 5.3
  >=10% | 11.3 | 13.2
  Unknown | 85.0 | 81.6

32. Primary Outcome: Percentage of Participants With Previous and Concurrent Disease at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
percentage of participants | 41.5 | 59.7

33. Primary Outcome: Percentage of Participants Who Received First-Line Endocrine Therapy at the Time of Local or Metastatic Progression
Description: as for outcome 10
Time Frame: At the time of Advanced or Metastatic Diagnosis (up to a maximum of 260 months, assessed retrospectively at Baseline)
Population: Efficacy population. Here number of participants analyzed were those who were available for the specified evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer
Number analyzed (Participants) | 124
percentage of participants | 24.2

34. Secondary Outcome: Percentage of Participants Who Maintained Bevacizumab Beyond the First Progressive Disease
Time Frame: as for outcome 18
Population: Efficacy population. Here number of participants were those who were available for this evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 104 | 53
percentage of participants | 25.0 | 17.0

35. Secondary Outcome: Percentage of Participants Who Received Induction Therapy in Combination With Bevacizumab
Time Frame: as for outcome 18
Population: Efficacy population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Number analyzed (Participants) | 135 | 67
percentage of participants | 99.3 | 98.5

ADVERSE EVENTS:
Time Frame: From inclusion (baseline) to 18 months
Groups:
- Bevacizumab: HR+ Breast Cancer: Participants with HER2- metastatic or locally advanced HR+ breast cancer, who received first-line bevacizumab in combination with chemotherapy for >=12 months and without disease progression for at least 12 months were included. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months. Bevacizumab treatment considering retrospectively and prospectively was approximately 61 months.
- Bevacizumab: TN Breast Cancer: Participants with HER2- metastatic or locally advanced TN breast cancer, who received first-line bevacizumab in combination with chemotherapy for >=12 months and without disease progression for at least 12 months were included. Participants who were alive at inclusion in the study, were prospectively followed for maximum of 18 months. Bevacizumab treatment considering retrospectively and prospectively was approximately 61 months.
Arm/Group | Bevacizumab: HR+ Breast Cancer | Bevacizumab: TN Breast Cancer
Serious Adverse Events (participants affected / at risk) | 10/150 | 4/77
Other Adverse Events (participants affected / at risk) | 7/150 | 9/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab: HR+ Breast Cancer (N=150) | Bevacizumab: TN Breast Cancer (N=77)
General physical health deterioration (General disorders) | 3 | 0
Death (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab: HR+ Breast Cancer (N=150) | Bevacizumab: TN Breast Cancer (N=77)
Asthenia (General disorders) | 4 | 5
Proteinuria (Renal and urinary disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.